CLINICAL TRIAL: NCT04661137
Title: A Phase 2B Study of Selinexor (KPT-330), in Combination With Carfilzomib, Daratumumab or Pomalidomide in Patients With Multiple Myeloma Relapsing on Current Therapy
Brief Title: A Study of Selinexor, in Combination With Carfilzomib, Daratumumab or Pomalidomide in Patients With Multiple Myeloma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment is paused pending an upcoming amendment
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020-0369; IST-318 (Other: Karyopharm)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Selinexor; KPT-330
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; carfilzomib; pomalidomide; daratumumab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Carfilzomib-containing Regimen (Experimental): Carfilzomib 56 mg/m2 on days 1, 8 and 15. Dexamethasone 20 mg if ≥ 75 years old and 40 mg if < 75 years old on days 1, 8, 15 and 22.
  Selinexor 80 mg on days 1, 8 and 15.
  Interventions: Drug: Selinexor 80 MG; Drug: Carfilzomib; Drug: Dexamethasone
- Pomalidomide-containing Regimen (Experimental): Pomalidomide 4 mg po daily for 21 days. Dexamethasone 20 mg if ≥ 75 years old and 40 mg if < 75 years old on days 1, 8, 15 and 22.
  Selinexor 60 mg on days 1, 8 and 15.
  Interventions: Drug: Selinexor 60 MG; Drug: Pomalidomide; Drug: Dexamethasone
- Exploratory/Daratumumab-containing Regimen (Experimental): Daratumumab on current schedule (16 mg/kg IV days 1, 8, 15 and 22 for cycles 1-2; days 1 and 15 for cycles 3-6; day 1 for cycle 7 and on).
  Dexamethasone 20 mg if ≥ 75 years old and 40 mg if < 75 years old on days 1, 8, 15 and 22.
  Selinexor 100 mg on days 1, 8, 15 and 22.
  Interventions: Drug: Selinexor 100 MG; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor 60 MG — Selinexor 60 mg PO on days 1, 8 and 15
  Other Names: KPT-330
  Arms: Pomalidomide-containing Regimen
Drug: Selinexor 80 MG — Selinexor 80 mg PO on days 1, 8 and 15
  Other Names: KPT-330
  Arms: Carfilzomib-containing Regimen
Drug: Selinexor 100 MG — Selinexor 100 mg PO on days 1, 8, 15 and 22
  Other Names: KPT-330
  Arms: Exploratory/Daratumumab-containing Regimen
Drug: Carfilzomib — 56 mg/m2 IV on days 1, 8 and 15
  Other Names: Kyprolis
  Arms: Carfilzomib-containing Regimen
Drug: Pomalidomide — 4 mg PO daily for 21 days
  Other Names: Pomalyst
  Arms: Pomalidomide-containing Regimen
Drug: Daratumumab — 16 mg/kg IV days 1, 8, 15 and 22 for cycles 1-2; days 1 and 15 for cycles 3-6; day 1 for cycle 7 and on
  Other Names: Darzalex
  Arms: Exploratory/Daratumumab-containing Regimen
Drug: Dexamethasone — 20 mg if ≥ 75 years old and 40 mg if < 75 years old on days 1, 8, 15 and 22
  Other Names: Dextenza, Ozurdex, Neofordex, others

SUMMARY:
This is a prospective, 2-arm (with an additional exploratory arm), open-label, multicenter study looking at the response rate of patients receiving selinexor (KPT-330), in combination with carfilzomib, daratumumab or pomalidomide.

Multiple Myeloma patients with documented disease progression or refractory disease while on current treatment with any carfilzomib-containing regimen (arm 1), any pomalidomide-containing regimen (arm 2) or any daratumumab-containing regimen (exploratory arm) will be included in the study. Patients will be assigned to the respective groups according to their current treatment. If a subject has received more than one of the above therapies, then assignment will be made at their physician's discretion (e.g treatment decision can be made based upon patient and physician preferred tolerance.).

Patients will receive treatment until progressive disease (PD), death, toxicity that cannot be managed by standard of care, or withdrawal, whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase 2b, two-arm, open-label, multicenter study of Sd (selinexor 100, 80 or 60 mg) in combination with carfilzomib, or pomalidomide in patients with MM previously treated with carfilzomib or pomalidomide respectively, and refractory to prior treatment. An additional exploratory arm will focus on patients treated with SD in combination with daratumumab.

This study will enroll approximately 96 patients overall (43 in each of the arms and 10 additional patients in the exploratory arm. Patients will be assigned to the respective arms based on their previous treatment.

Patients who are relapsed or refractory to their current carfilzomib-based regimen will be enrolled on Arm 1 and will receive the following treatment regimen on a 28-day cycle:

Carfilzomib 56 mg/m2 on days 1, 8 and 15. They will also receive dexamethasone 40 mg (or 20 mg if patient is ≥ 75 years old) once weekly and Selinexor 80 mg on days 1, 8 and 15.

Patients who are relapsed or refractory to their current pomalidomide-based regimen will be enrolled on Arm 2 and will receive the following treatment regimen on a 28-day cycle:

Pomalidomide 4 mg po daily for 21 days combined with Dexamethasone 40 mg (or 20 mg if patient is ≥ 75 years old) once weekly and Selinexor 60 mg days 1, 8 and 15.

For arms 1 and 2, 13 patients will be accrued in each arm in the first stage. If there are 3 or fewer responses in these 13 patients, the study will be stopped. Otherwise, 30 additional patients will be accrued for a total of 43 (in each arm).

Finally, in the exploratory arm, we will enroll up to 10 patients who are relapsed or refractory to their current daratumumab-based regimen. Patients enrolled on the exploratory arm will receive the following treatment regimen on a 28-day cycle:

Daratumumab on current schedule (16 mg/kg IV days 1,8,15,22 for cycles 1-2; days 1 and 15 for cycles 3-6; day 1 for cycle 7 and on) combined with Dexamethasone 40 mg once weekly (or 20 mg if patient is ≥ 75 years old) and Selinexor 100 mg once weekly.

The Investigator may remove a patient from study treatment using criteria described in Section 10.2. Patients may decide to discontinue study treatment for any reason. Patients who elect to discontinue study treatment should be encouraged to continue in the study so that follow-up information on disease progression, other antineoplastic therapy, symptoms and survival status may be obtained. However, patients may elect to withdraw consent and decline further participation in the trial at any time.

The Investigator must determine the primary reason for a patient's discontinuation of study treatment and record this information on the electronic case report form (eCRF). Patients who are prematurely withdrawn from study treatment are not eligible to re-initiate study treatment on this protocol at a later date.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of informed consent.
2. Histologically confirmed MM and evidence of disease progression while on one of the below MM regimens:

   * Arm 1: Refractory to or disease progression while on a carfilzomib-containing regimen
   * Arm 2: Refractory to or disease progression while on a pomalidomide-containing regimen
   * Exploratory Arm: Refractory to or disease progression while on a daratumumab-containing regimen
3. Measurable disease as defined: Serum M-protein ≥ 0.5 g/dL; urine M-protein excretion at least 200 mg/24h; serum FLC ≥ 100 mg/L, provided that FLC is abnormal; if serum protein electrophoresis is felt to be unreliable for routine M-protein measurement (i.e. IgA MM) then quantitative Ig levels by nephelometry or turbidometry are acceptable; for non-secretory disease, bone marrow plasma cells ≥ 20% or a biopsy-proven target lesion by PET/CT or MRI is acceptable
4. Documented evidence of disease progression (by IMWG criteria) or refractory disease on the current treatment as defined as:

   * Achieving SD or less for ≥ 1 cycle during treatment with regimens stated in #2 (i.e. relapsed) OR
   * <25% response (i.e. never achieved MR) or PD during or within 60 days from the end-of most recent MM regimen as listed in #2 (i.e. refractory).
5. Any non-hematological toxicities (except for peripheral neuropathy) that patients experienced from treatments in previous regimens have resolved to Grade 2 or less by Cycle 1 Day 1.
6. ECOG 2 or less
7. Adequate hepatic function within 28 days prior to C1D1:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to <2 × ULN.
8. Adequate renal function within 28 days prior to C1D1 as determined by estimated creatinine clearance of ≥ 30 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female (Cockcroft 1976).
9. Adequate hematopoietic function within 7 days prior to C1D1: total white blood cell (WBC) count ≥1500/mm3, absolute neutrophil count ≥1000/mm3, hemoglobin ≥8.5 g/dL and platelet count ≥75,000/mm3 (patients for whom <50% of bone marrow nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of bone marrow nucleated cells are plasma cells).

   1. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.
   2. Patients must have:

      * At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and
      * At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment.

   However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
10. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

  1. Smoldering MM
  2. Radiation therapy, chemotherapy or immunotherapy other than above stated regimens in #2 ≤2 weeks prior to C1D1. Patients on long-term glucocorticosteroids during screening do not require a washout period. Prior RT is permitted for treatment of fractures or to prevent fractures as well as for pain management.
  3. Active graft versus host disease after allogeneic stem cell transplant.
  4. Life expectancy <3 months.
  5. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus ribonucleic acid (RNA) or hepatitis B virus surface antigen.
  6. Has any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
  7. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
  8. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
  9. Pregnant or breastfeeding females.
  10. Body surface area (BSA) <1.4 m2 at baseline, calculated by the Dubois (Dubois 1916) or Mosteller (Mosteller 1987) method.
  11. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
  12. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Comprehensive Cancer Network® (NCCN) Clinical Practice Guidelines in Oncology (CPGO) (NCCN CPGO) for antiemesis and anorexia/cachexia (palliative care).
  13. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
  14. Contraindication to any of the required concomitant drugs or supportive treatments.
  15. Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of patients receiving selinexor with carfilzomib and dexamethasone (Arm 1) | 30 Months
  ORR will include patients who experience partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR), based on International Myeloma Working Group (IMWG) response criteria (Kumar 2016)
Overall Response Rate (ORR) of patients receiving selinexor with pomalidomide and dexamethasone (Arm 2) | 30 Months
  ORR will include patients who experience partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR), based on International Myeloma Working Group (IMWG) response criteria (Kumar 2016)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 30 Months
  Duration from start of study treatment to PD or death [regardless of cause], whichever comes first
Overall Survival (OS) | 30 Months
  Duration from start of study treatment to death
MRD Negativity | 30 Months
  Rate of achievement of minimal residual disease (MRD) by multiparametric flow cytometry
Incidence of Adverse Events [Safety and Tolerability] using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), v 4.03. | 30 Months
  Incidence of Adverse Events [Safety and Tolerability] using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), v 4.03.
Time To Next Treatment (TTNT) | 30 Months
  Duration from start of study treatment to next treament

OTHER OUTCOMES:
Overall Response Rate (ORR) of patients receiving selinexor with daratumumab and dexamethasone | 30 Months
  ORR will include patients who experience partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR), based on International Myeloma Working Group (IMWG) response criteria (Kumar 2016)
Gut Microbiome analysis | 30 Months
  To identify intestinal microbiota associated biomarkers that predict response and risk for development of treatment-related toxicities at baseline, on-treatment, post-treatment and relapse.
Immune cell subset analyses | 30 Months
  Changes from baseline in immune cell subsets in peripheral blood mononuclear and bone marrow mononuclear cells will be monitored.
Analyses of cytokine markers | 30 Months
  Cytokines will be quantified in plasma samples by multiplex ELISA and other readout assays.
Analyses of chemokine markers | 30 Months
  Chemokines will be quantified in plasma samples by multiplex ELISA and other readout assays.
Analyses of inflammatory/anti-inflammatory markers | 30 Months
  Inflammation/anti-inflammation markers will be quantified in plasma samples by multiplex ELISA and other readout assays.
Analyses of bacterial translocation markers | 30 Months
  Bacterial translocation markers will be quantified in plasma samples by multiplex ELISA and other readout assays.
Basic peripheral blood laboratory variables: Lymphocytes | 30 Months
  Basic peripheral blood laboratory value of absolute and relative lymphocytes obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: Eosinophils | 30 Months
  Basic peripheral blood laboratory value of absolute and relative eosinophils obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: Monocytes | 30 Months
  Basic peripheral blood laboratory value of absolute and relative monocytes obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: Neutrophils | 30 Months
  Basic peripheral blood laboratory value of absolute and relative neutrophils obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: Basophils | 30 Months
  Basic peripheral blood laboratory value of absolute and relative basophils obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: LDH | 30 Months
  Basic peripheral blood laboratory value of LDH obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Basic peripheral blood laboratory variables: Neutrophil-to-lymphocyte ratio (NLR) | 30 Months
  Basic peripheral blood laboratory value of absolute neutrophil-to-lymphocyte ratio (NLR) obtained in routine clinical care will be evaluated prior to treatment, on-treatment, post-treatment, relapse and at development of severe AE (>3 score).
Analyses of genetic profiles | 30 Months
  Exploratory analysis to identify molecular genomic determinants of response or resistance to selinexor in the treatment combinations to define biomarkers
Analyses of markers of de novo or acquired resistance to treatment | 30 Months
  Exploratory analysis to identify mechanisms of de novo or acquired resistance to selinexor in combination with carfilzomib, pomalidomide or daratumumab.

CONTACTS AND LOCATIONS:
Overall Officials: Noa Biran, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Du Bois D, Du Bois EF. A formula to estimate the approximate surface area if height and weight be known. 1916. Nutrition. 1989 Sep-Oct;5(5):303-11; discussion 312-3. No abstract available. PMID 2520314
- [Background] Mosteller RD. Simplified calculation of body-surface area. N Engl J Med. 1987 Oct 22;317(17):1098. doi: 10.1056/NEJM198710223171717. No abstract available. PMID 3657876
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Fridericia L. Die Systolendauer im elektrokardiogramm bei normalen menschen und bei herzkranken. [The duration of systole in the electrocardiogram of normal subjects and of patients with heart disease.]. Acta Medica Scandinavica. 1920;53:469-86.
- [Background] Bahlis N, Chen C, Sebag M et al. A Phase 1B/2 Study of Selinexor in combination with backbone therapies for treatment of relapsed/refractory multiple myeloma. EHA Learning Center. Abstract P277. June 10, 2016.
- [Background] Jakubowiak A, Jasielec J, Rosenbaum CA et al. Final Results of Phase 1 MMRC Trial of Selinexor, Carfilzomib, and Dexamethasone in Relapsed/Refractory MM. Blood 2016. 128;973.
- [Background] Chari A, et al. Results of the Pivotal STORM Study (Part 2) in Penta-Refractory Multiple Myeloma (MM): Deep and Durable Responses with Oral Selinexor Plus low dose Dexamethasone in Patients with Penta-Refractory MM. Blood. 2018. ASH Abstract 598.
- [Background] Gasparetto C, et al. Deep and Durable Respones with Selinexor, Daratumumab and Dexamethasone (SDd) in Patients with MM Previously Exposed to Proteasome Inhibitors and Immunomodulatory Drugs: Results of the Phase 1B Study of SDd. Blood 2018. ASH Abstract 599.
- [Background] Gasparetteo C, Lipe B, Tuchman S, et al. Once weekly selinexor, carfilzomib, and dexamethasone (SKd) in patients with relapsed/refractory multiple myeloma (MM). Poster presented at the 2020 American Society of Clinical Oncology Virtual Annual Meeting. J Clin Oncol 38:2020 (suppl; abstr 8530)
- [Background] Chen CI, Bahlis N, Gasparetto C, et al. Selinexor, pomalidomide, and dexamethasone (SPd) in patients with relapsed or refractory multiple myeloma. Presented at: American Society of Hematology Annual Meeting; Orlando, Florida. December 6-10, 2019.
- [Background] Gasparetto C, Lentzsch S, Schiller GJ et al). Selinexor, daratumumab and dexamethasone in patients with relapsed/refractory multiple myeloma (MM). Poster presented at the 2020 American Society of Oncology Virtual Annual Meeting. J Clin Oncol 38: 2020 (Suppl abstr 8510)